CLINICAL TRIAL: NCT00891449
Title: Countermeasure and Functional Testing Study (CFT-70)
Brief Title: Space Flight Simulation to Study Effects of Micro-gravity Through Bed Rest
Acronym: FAP
Status: Completed | Type: Observational
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SA-06-2770
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Weightlessness
Keywords: space flight simulation study; medical research study; bed rest; microgravity; weightlessness; The effects of long duration microgravity on humans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Space flight simulation study to study effects of microgravity through bedrest coupled with flight exercise counter-measures.

DETAILED DESCRIPTION:
Flight Analogs/Bed Rest Research Project (FA/BRRP) provides NASA with a ground-based research platform to complement space research. By mimicking on Earth the conditions of weightlessness experienced by the human body in space, NASA can test and refine scientific theories and procedures to develop countermeasures to protect humans from the effects of the space travel. The use of ground analogs, such as bed rest, are essential because access to the resources required to conduct studies in space is very limited, and the expense of studies significantly greater than those conducted using flight analogs. Future space exploration will challenge NASA to answer many critical questions about how humans can live and work for extended missions away from Earth.

Flight analog testing is critical to NASA to validate countermeasures, given the few opportunities to use flight platforms as the Shuttle retires; also, the US has only 1-2 International Space Station (ISS) crewmembers per Expedition. The Flight Analogs/Bed Rest Research Project is one way NASA will devise ways to ensure astronaut safety and productivity on extended missions to the moon and Mars.

In the Flight Analogs Project (FAP), volunteers spend many days in a controlled research environment in the Flight Analog Research Unit (FARU) in Galveston, TX. In the current campaigns, volunteers will undergo three phases in the bedrest projects: 1) pre-bedrest baseline testing, 2) a bedrest phase, and 3) the recovery period. Bed rest results in many physiologic changes similar to those seen in astronauts. Pre bed rest is used to gather baseline data against which the bed-rest phase data will be compared. Researchers then monitor how the volunteers' bodies change over the course of the study and how quickly they recover once they are allowed to resume normal activities. Post bed rest is used to monitor recovery from bed rest. In longer campaigns, return to the unit for follow-up testing may be requested after 1, 3, 6, and/or 12 months.

THE COUNTERMEASURE AND FUNCTIONAL TESTING STUDY (CFT) will test the effectiveness of exercise on loss of muscle, bone and cardiovascular function. Participants will perform an exercise program in a system called the standalone Zero Gravity Locomotion Simulator (sZLS), a "vertical treadmill" that removes the weight from the long axis of the body to simulate exercise as it is done in space. Resistance (weight lifting) exercise will be performed on special weight machines. Before and after 70 days of bedrest, participants will be tested on a corresponding set of physiological measures. Specific exercises and intensities are rotated such that each workout is different, with some days being heavier and some lighter. Results of the study will help understand which mission tasks might be affected by changes in physiology during space flight and design countermeasures to prevent or minimize impairment to these physiological systems

The ALTERNATE COMPRESSION GARMENT STUDY (ACG) will determine effectiveness of compression garments on regulating blood pressure and other body systems after extended periods of head-down bed rest. Participants in the experimental group will wear custom-fit compression garments and undergo evaluation on their response to an upright tilt test and a corresponding set of physiological measures before and after 14 days of bed rest. These participants will be compared to another group of participants who did not wear the compression garments. Results of the study will help scientists determine the time it takes for the cardiovascular system to re-adapt to upright posture, determine whether wearing compression garments during recovery is necessary to protect against dizziness and loss of consciousness often experienced after space missions, and determine the effect of wearing custom fit compression garments on the amount of time needed to readjust to a normal, upright posture.

ELIGIBILITY:
Inclusion Criteria:

* US Citizen
* Must be able to pass physical

Exclusion Criteria:

* tobacco use
* menopausal
* prescription drug use
* food allergies
* joint injuries
* Thrombosis
* Reflux
* High blood pressure
* Diabetes

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ronita L Cromwell, Ph.D., Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Dillon EL, Soman KV, Wiktorowicz JE, Sur R, Jupiter D, Danesi CP, Randolph KM, Gilkison CR, Durham WJ, Urban RJ, Sheffield-Moore M. Proteomic investigation of human skeletal muscle before and after 70 days of head down bed rest with or without exercise and testosterone countermeasures. PLoS One. 2019 Jun 13;14(6):e0217690. doi: 10.1371/journal.pone.0217690. eCollection 2019. PMID 31194764
- See also: Popular Science: Pillownauts Stay in Bed for the Sake of Science — http://www.popsci.com/military-aviation-amp-space/article/2009-06/pillownaut-stays-bed-sake-science